CLINICAL TRIAL: NCT00166413
Title: A Phase II Trial of CC-5013 in Patients With Primary Systemic Amyloidosis
Brief Title: Efficacy of CC-5013 (Revlimid or Lenalidomide) in Patients With Primary Systemic Amyloidosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Angela Dispenzieri, M.D., Mayo Clinic Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1105-04; MC0484 (Other: Mayo Clinic Cancer Center); 1105-04 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2011-05-06 (Estimated); Status verified 2011-05

CONDITIONS: Amyloidosis
MeSH Terms: conditions — Amyloidosis | interventions — Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CC5013 (Experimental): Assess the proportion of confirmed hematologic responses (HCR, HPR) resulting from treatment with CC5013 after 3 months in patients with primary systemic amyloidosis.
  Interventions: Drug: CC-5013

INTERVENTIONS:
Drug: CC-5013 — 40 mg/day orally on days 1-4 and 15-18 of each 28-day cycle
  Other Names: amino substituted analog of thalidomide

SUMMARY:
Patients with primary systemic amyloidosis will be treated with CC-5013 (lenalidomide; Revlimid) as a single agent for 3 months. If their disease worsens or does not improve during that time frame dexamethasone will be added to the treatment program.

ELIGIBILITY:
1. Histochemical diagnosis of amyloidosis as based on detection by polarizing microscopy of green birefringent material in Congo red-stained tissue specimens and immunohistochemical proof of AL
2. Measurable disease of AL amyloidosis as defined by one of the following:

   * Serum monoclonal protein >=1.0 g by protein electrophoresis
   * >200 mg of monoclonal protein in the urine on 24 hour electrophoresis
   * Serum immunoglobulin free light chain & >=10 mg/dL AND abnormal serum immunoglobulin kappa to lambda free light chain ratio
3. ECOG performance status (PS) 0, 1, 2, or 3
4. >=18 years of age
5. The following laboratory values obtained <=14 days prior to registration:

   * Creatinine < = 3 mg/dL
   * Absolute neutrophil count >=1000/microliter
   * Platelet >=75000/microliter
   * Hemoglobin > = 8.0 g/dL
6. Symptomatic organ involvement with amyloid to justify therapy. This could include liver involvement, cardiac involvement, renal involvement, peripheral neuropathy grade 1, or soft tissue involvement. Must have more than purpura or carpal tunnel syndrome
7. Previously treated or untreated. No limit to prior therapy provided there is adequate residual organ function
8. Ability to provide informed consent
9. Anticipated life expectancy of at least 3 months
10. None of the following:

    * Pregnant women or women of reproductive ability who are unwilling to use effective contraception
    * Nursing women
    * Men who are unwilling to use a condom (even if they have undergone a prior vasectomy) while having intercourse with any woman, while taking the drug and for 4 weeks after stopping treatment
    * Myelosuppressive chemotherapy < 4 weeks prior to registration
    * Concomitant high dose corticosteroids
    * Grade 2 (or higher) peripheral neuropathy
    * Uncontrolled infection
    * Clinically overt multiple myeloma
    * Active malignancy
    * Prior hypersensitivity reaction to Thalidomide
    * Syncope within the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2005-04; Primary Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the hematologic response rate of CC-5013 in patients with primary systemic amyloidosis | 12 months

SECONDARY OUTCOMES:
Toxicity of single agent CC-5013 and combination CC-5013 and dexamethasone | 12 months
Hematologic response rate of CC-5013 and dexamethasone | 12 months
Organ response of CC-5013 and the CC-5013 dexamethasone combination | 12 months
Time to progression | 5 years
Survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Angela Dispenzieri, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States